CLINICAL TRIAL: NCT05267509
Title: Identification of the Immuno Suppressive Characteristics of Glioma Patients by an Integrated Radio-immunological Approach
Brief Title: An Integrated Radio-immunological Approach
Acronym: IMMUNO-IMAGING
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other); Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/27
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Glioma, Malignant
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Glioma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The most aggressive primary brain tumors in adults, glioblastomas, are characterized by a profound local and systemic immune suppression. During tumor progression, the infiltration of inflammatory leukocytes, especially of myeloid origin, endowed with immunosuppressive function is observed. Aim of this study is to evaluate myeloid cell infiltrate and iron metabolism in tumor-associated macrophages by combining a multimodal MRI imaging technique with immunophenotyping of the tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* All patients with histologic confirmation of malignant glioma
* Patients must be age >= 18 years
* Patients must be able to obtain an MRI scan with gadolinium contrast
* Patients must sign informed consent indicating that they are aware of the investigational nature of this study:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologic confirmation of malignant glioma
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate leukocyte/myeloid cell-infiltrate in gliomas by using a multimodal PET/MRI imaging technique | 24 months
  apply iron-sensitive MRI sequences in glioma patients to identify macrophage iron deposits as biomarker of in vivo immune suppression, and correlate these findings with 5-Ala intraoperative data and analysis of MG and BMDM infiltration.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Mandruzzato, PhD, Principal Investigator — Istituto Oncologico Veneto IOV-IRCCS
Locations (2):
- Italy (2):
  - University Hospital, Florence
  - University Hospital, Padua